CLINICAL TRIAL: NCT04701515
Title: Cardiovascular Manifestations of COVID-19
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Methodist Health System (Other)
Responsible Party: Sponsor
Other Study IDs: 030.CVS.2020.D
Record Dates: First submitted 2020-09-22; First posted 2021-01-08 (Actual); Last update posted 2023-07-12 (Actual); Status verified 2023-07

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Retrospective Cohort: Review electronic medical records of de-identified patients that tested positive for COVID-19 (using a PCR test) at Methodist Dallas Medical Center (MDMC) from June 2020 until December 2022
  Interventions: Other: Chart review

INTERVENTIONS:
Other: Chart review — Chart review

SUMMARY:
Electronic medical record review of de-identified patients who tested positive for COVID-19 (using a PCR test) at Methodist Dallas Medical Center (MDMC) from June 2020 until the date of IRB approval. Data will be collected on de-identified patients that test positive for COVID-19 (using a PCR test) at MDMC from the date of IRB approval until December 2022. Disclaimer: Any cost associated with the procedures stated herein will be billed directly to you or to your insurance (as applicable)

DETAILED DESCRIPTION:
Electronic medical record review of de-identified patients who tested positive for COVID-19 (using a PCR test) at Methodist Dallas Medical Center (MDMC) from June 2020 until the date of IRB approval. Data will be collected on de-identified patients that test positive for COVID-19 (using a PCR test) at MDMC from the date of IRB approval until December 2022. Variables include patient baseline characteristics, patient presentation, imaging and labs. Disclaimer: Any cost associated with the procedures stated herein will be billed directly to you or to your insurance (as applicable)

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized patient
* Adult over 18 years
* Positive COVID-19 PCR Test

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients that test positive for COVID-19 (using a PCR test) at MDMC
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-03-21 (Actual); Primary Completion 2024-05-21 (Estimated); Study Completion 2024-05-21 (Estimated)

PRIMARY OUTCOMES:
Heart failure | March 2020 - June 2021
  Presence or absence
Tamponade | March 2020 - June 2021
  Presence or absence
Pericardial Effusion | March 2020 - June 2021
  Presence or absence
Myocarditis | March 2020 - June 2021
  Presence or absence
Pericarditis | March 2020 - June 2021
  Presence or absence
Arrythmias | March 2020 - June 2021
  Presence or absence
Troponin I | March 2020 - June 2021
  Level
N-terminal prohormone BNP | March 2020 - June 2021
  Level

SECONDARY OUTCOMES:
Stroke | March 2020 - June 2021
  Presence or absence
Myocardial infarction | March 2020 - June 2021
  Type
Shock | March 2020 - June 2021
  Presence or absence
Deep venous thrombosis | March 2020 - June 2021
  Presence or absence
Discharge disposition | March 2020 - June 2021
  Location
Primary diagnosis | March 2020 - June 2021
  Diagnosis upon discharge
Rate of ICU admission/transfer | March 2020 - June 2021
  Rates
Total hospital length of stay | March 2020 - June 2021
  Number of Days
ICU length of stay | March 2020 - June 2021
  Number of Days
Percentage of patients in cohort that had EKG testing or Echocardiography | March 2020 - June 2021
  Percentage

CONTACTS AND LOCATIONS:
Overall Officials: Manavjot Sidhu, MD, Principal Investigator — Methodist Health System
Locations (1):
- Methodist Dallas Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No